CLINICAL TRIAL: NCT04009382
Title: Modulation Effects of Baduanjin Mind-body Exercise on Subjective Cognitive Decline
Brief Title: Modulation Effects of Baduanjin Exercise on Subjective Cognitive Decline
Acronym: BDJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018P001997
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin (Experimental): This group will participate in the Baduanjin exercise intervention for 24 weeks (three times/week for the first three months and two times/week for the last three months).
  Interventions: Other: Baduanjin Exercise
- Cognitive Fitness Program (Active Comparator): This group will participate in the Cognitive Fitness Program intervention for 24 weeks (three times/week for the first three months and two times/week for the last three months).
  Interventions: Other: Cognitive Fitness Program

INTERVENTIONS:
Other: Baduanjin Exercise — Subjects will participate in Baduanjin, a simple mind-body exercise, for 24 weeks.
  Arms: Baduanjin
Other: Cognitive Fitness Program — Subjects will complete paper puzzles (Sudoku, crosswords, etc.) for 24 weeks.
  Arms: Cognitive Fitness Program

SUMMARY:
The aim of this study is to investigate the modulation effects of Baduanjin (BDJ), a simple and innovative mind-body exercise, on cognitive function, resting state functional connectivity, and brain morphometry in individuals with subjective cognitive decline (SCD). The results obtained will provide novel insights for improving the prevention of age-related cognitive decline and Alzheimer's disease.

DETAILED DESCRIPTION:
Subjective cognitive decline (SCD), the self-reported perception of memory or cognitive problems, is receiving increasing attention as a risk factor for the development of Alzheimer's disease (AD). Since SCD manifests before the onset of clinical impairment, it might be the optimal stage/window of time at which to intervene with preventative therapies for AD and age-related dementia before the progressive neurological loss and irreversible cognitive impairment.

Recently, mind-body interventions have demonstrated their potential in preventing cognitive decline. Nevertheless, these mind-body therapies encompass a family of complex practices, each with different characteristics and focus. Therefore, they may be associated with different mechanisms and treatment effects. Baduanjin (BDJ) is an innovative and simple mind-body exercise consisting of eight simple movements that can be easily practiced at home with video guidance, thereby making it a more suitable option for older adults with cognitive decline than other more complex exercises.

We believe that this study will 1) significantly improve the prevention of MCI and AD and directly benefit patients suffering from these highly prevalent disorders, 2) enhance the investigators' understandings of the neurobiology through which mind-body interventions affect cognition and health, and 3) advance the investigators' understandings of the pathophysiology and development of SCD, AD, and age-related dementia.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 80 years old
* Self-reported experience of persistent decline in memory compared with a previous state (within the past 5 years), which was further confirmed by informants
* Concerns regarding memory problems
* Mini-Mental State Examination, Second Edition (MMSE-2) scores within the normal range
* Montreal Cognitive Assessment scores within the normal range (adjusted for age, sex, and education)
* Clinical Dementia Rating score of 0 (no memory loss or slight, inconsistent forgetfulness)

Exclusion Criteria:

* Unable to speak or read English
* Diagnosis of depression
* Other diseases that cause cognitive decline (e.g., traumatic brain injury, stroke, neurodegenerative diseases, brain tumor, Parkinson disease, encephalitis or epilepsy, thyroid dysfunction, severe anemia, syphilis)
* History of psychosis or congenital mental growth retardation
* Any delayed recall index greater than 1.5 SD below average on the California Verbal Learning Test, Second Edition
* Failing the Memory items on the MMSE-2 and MDRS-2, as well as the CVLT-II criterion
* Inability to participate in a 6-month intervention with a 3-month follow-up
* Any item = 0 on the Lawton-Brody Instrumental Activities of Daily Living Scale for cognitive reasons
* No available informant
* Previous diagnosis of MCI, AD, or other age-related dementia
* Previous Baduanjin experience

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Alzheimer Disease Cooperative Study- Preclinical Alzheimer (ADCS-PACC) Cognitive Composite | baseline, 3, 6, 9 months
  The ADCS-PACC is a composite of well-validated neuropsychological tests that were selected specifically due to their sensitivity in tracking the earliest evidence of decline from normal to subtly abnormal cognitive performance.
Functional connectivity of hippocampus and DLPFC | baseline, 3, 6 months
  Resting state functional connectivity of the hippocampus and dorsolateral prefrontal cortex (DLPFC) based on resting state functional magnetic resonance imaging (fMRI) data will be used.

SECONDARY OUTCOMES:
Everyday Cognition -Subject/Self Report Form (ECog-self report and informant) | baseline, 3, 6, 9 months
  The Ecog was developed to 1) measure relatively mild functional changes that may predate loss of independence in major activities of daily living; and 2) assess functional abilities that are clearly linked to specific cognitive abilities.
Patient Reported Outcomes Measurement Information System 29 (PROMIS-29) | baseline, 3, 6, 9 months
  PROMIS-29 will be used to assess physical function, depression, anxiety, fatigue, sleep, social activity and pain in the past 7 days.
Brain morphometry | baseline, 3, 6 months
  The imaging endpoint is to assess brain grey matter volume changes using before and after BDJ exercise and magnetic resonance imaging (MRI).
Blood markers | baseline, 3, 6, 9 months
  Circulating markers, such as C reactive protein, proinflammatory cytokine IL-6, and BDNF will be measured to investigate the modulation effect of Baduanjin.
Heart rate variability | baseline, 3, 6, 9 months
  The secondary endpoints include measuring low frequency, high frequency, and LF to HF ratio (LF/HF) of heart rate variability as measured by ECG.
Beck Anxiety Inventory (BAI) | baseline, 3, 6, 9 months
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety in children and adults
Symbol Digit Modalities Test (SDMT) | baseline, 3, 6, 9 months
  This is an oral version of the Digit Symbol Substitution Test
The Stroop Color and Word Test (SCWT) | baseline, 3, 6, 9 months
  This is a test to assess executive functions, the ability to inhibit cognitive interference, attention, processing speed, and cognitive flexibility.
Trail-making Test A and B | baseline, 3, 6, 9 months
  This is a test of speeded visual search, vigilance, and set-shifting.
Controlled Oral Word Association Test, Category Fluency and Category Switching | baseline, 3, 6, 9 months
  These are tests of rapid word retrieval, cognitive flexibility, and semantic access/semantic network integrity.
Patient Reported Outcomes Measurement Information System - Cognition Function and ability subset | baseline, 3, 6, 9 months
  The PROMIS Cognitive Function and Cognitive Function Abilities Subset item banks assess patient-perceived cognitive deficits
The California Verbal Learning Test-II (CVLT-II) | baseline, 3, 6, 9 months
  CVLT-II is a comprehensive assessment of verbal learning and memory available for older adolescents and adults.
Modified Brief Pain Inventory (BPI) | baseline, 3, 6, 9 months
  The BPI is a 15-item questionnaire rating pain location, intensity, relief, quality, and pain-related quality of life.
Brief Quantitative Sensory Testing (QST) | baseline, 3, 6, 9 months
  QST will include mechanical and heat pain threshold and tolerance measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States